CLINICAL TRIAL: NCT06004752
Title: A Single-center, Single-arm, Prospective Clinical Study on the Efficacy and Safety of Cyclosporine Combined With Avatrombopag in the Treatment of Non-severe Aplastic Anemia in the Elderly
Brief Title: Efficacy and Safety of CsA+AVA in the Treatment of NSAA in the Elderly
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avatrombopag-2
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclosporine; avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Cyclosporine: 3mg/kg/d 3-5mg/kg bid was administered to maintain the trough concentration at 100-200 μg/ml;
  Avatrombopag: The dosage was 40~60mg orally, once a day, and the dosage was adjusted according to the subject's platelet count. The drug was administered for 24 weeks (6 months).
  Interventions: Drug: Ciclosporin; Drug: Avatrombopag

INTERVENTIONS:
Drug: Ciclosporin — Cyclosporine was taken orally at 3-5mg/kg bid was administered to maintain the trough concentration at 100-200 μg/ml
Drug: Avatrombopag — Avatrombopag was administrated at 40 mg/d and increased by 20 mg/d during the biweekly follow-up if platelet was not 20 × 109/L higher than baseline. AVA dose was gradually reduced if PLT ≥ 150 × 109/L. The maximum dose was 60 mg/d, while the minimum was 20 mg/week.

SUMMARY:
For elderly patients who cannot tolerate anti-thymocyte globulin (ATG) treatment, the addition of avatrombopag (AVA), which has a slight adverse reaction, can theoretically improve the hematological response rate in elderly patients with non-severe aplastic anemia (NSAA) without significantly increasing adverse reactions. Based on this, this study treated NSAA patients older than 60 with AVA combined with CsA to evaluate the hematological response rate and safety of AVA in the elderly who could not tolerate ATG therapy.

DETAILED DESCRIPTION:
Aplastic anemia (AA) can be divided into severe AA (SAA) and non-severe AA (NSAA), according to the severity of the disease. Anti-thymocyte globulin (ATG) in combination with CsA is the most typical combined immunosuppressive therapy regimen. For elderly patients who cannot tolerate anti-thymocyte globulin (ATG) treatment, the addition of avatrombopag, which has a slight adverse reaction, can theoretically improve the hematological response rate in elderly patients with NSAA without significantly increasing adverse reactions. Based on this, this study treated NSAA patients older than 60 with AVA combined with CsA to evaluate the hematological response rate and safety of AVA in the elderly who could not tolerate ATG therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients with well-defined NSAA anemia who meet the diagnostic criteria for aplastic anemia (AA) but do not meet the diagnostic criteria for severe aplastic anemia (SAA).
2. Age 60 years or older, male or female.
3. Able to swallow or administer orally.
4. Intolerant or refused anti-thymocyte globulin treatment

6. No previous treatment with cyclosporine, tacrolimus or hormones or treatment for less than 1 month.

7. No prior treatment with thrombopoietin (TPO) receptor agonists (including eltrombopag, herombopag, romiplostim, etc.) 8. Informed consent must be signed before the start of all specific research procedures. Considering the patient's condition, if the patient's signature is not conducive to the treatment of the disease, the informed consent shall be signed by the patient's immediate family.

Exclusion Criteria:

1. Known congenital AA (such as Fanconi anemia) and other causes of pancytopenia and hematological bone marrow disorders;
2. With paroxysmal nocturnal hemoglobinuria (PNH) clone ≥ 50%
3. With a history of hematopoietic stem cell transplantation.
4. History of thrombosis
5. Patients with underlying cancer who also have malignant tumors or are receiving immunosuppressive therapy.
6. Baseline creatine levels greater than twice of the upper limit of normal (ULN) and/or alanine aminotransferase (ALT) greater than 2.5 times of the ULN;
7. Serious heart, liver and kidney disease.
8. With uncontrolled bleeding and/or infection after standard treatment.
9. Participants considered unsuitable for inclusion by the researchers.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
ORR at 6 Months | 6 months
  Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
Changes in Haemoglobin in the Absence of Red Blood Cells Transfusion | 6 months
  The change in hematology values ( haemoglobin) were evaluated
Changes in Platelet in the Absence of Platelet Transfusion | 6 months
  The change in hematology values (platelet) were evaluated
Percentage of patients with clonal evolution to myelodysplasia, PNH, acute leukemia | 12 months
  Clonal evolution to myelodysplasia is defined as a new marrow cytogenic abnormality with or without characteristic dysplastic marrow findings. Evolution to leukemia is defined as greater than 20% peripheral blood and/or marrow blasts. Evolution to paroxysmal nocturnal hemoglobinuria (PNH) is defined as a clone at baseline < 10% that rose to greater than 50% on study.
ORR at 1, 2, 3 Months and at the end of follow-up | 1, 2, 3 Months, last follow-up
  Overall Response Rate (ORR) Defined as the Number of Participants Who Met the Criteria of Either Complete Response (CR) or Partial Response (PR)
Relapse rate | 6 months, last follow-up
  Relapse was defined as a substantial or progressive decline in at least one blood lineage counts of the responders that required the reinitiation or augmentation of AVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data would be accepted upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: always
Access Criteria: email request